CLINICAL TRIAL: NCT03033069
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo- and Active-controlled Trial of Brexpiprazole (1 - 3 mg/Day) as Monotherapy or as Combination Therapy in the Treatment of Adults With Post-traumatic Stress Disorder
Brief Title: A Study of Flexible Dose Brexpiprazole as Monotherapy or Combination Therapy in the Treatment of Adults With Post-traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-201-00061
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — brexpiprazole; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Brexpiprazole + Sertraline (Experimental): Participants were administered oral brexpiprazole initial dose of 0.5 milligram (mg)/day plus sertraline initial dose of 50 mg/day. The dose was up titrated to brexpiprazole maximum dose of 3 mg/day and sertraline maximum dose of 200 mg/day and continued thereafter up to Week 12 based on efficacy and tolerability. No dose reductions were allowed after Week 6 and no dose increments were allowed after Week 4. Participants also received sertraline matching placebo based on dose titration/adjustment up to Week 12.
  Interventions: Drug: Brexpiprazole; Drug: Sertraline; Drug: Sertraline Matching Placebo
- Brexpiprazole (Experimental): Participants were administered oral brexpiprazole initial dose of 0.5 mg/day The dose was up titrated to brexpiprazole maximum dose of 3 mg/day and continued thereafter up to Week 12 based on efficacy and tolerability. No dose reductions were allowed after Week 6 and no dose increments were allowed after Week 4. Participants also received sertraline matching placebo up to Week 12.
  Interventions: Drug: Brexpiprazole; Drug: Sertraline Matching Placebo
- Sertraline (Active Comparator): Participants were administered oral sertraline initial dose of 50 mg/day. The dose was up titrated to sertraline maximum dose of 200 mg/day and continued thereafter up to Week 12 based on efficacy and tolerability. No dose reductions were allowed after Week 6 and no dose increments were allowed after Week 4. Participants also received brexpiprazole matching placebo and sertraline matching placebo based on dose titration/adjustment up to Week 12.
  Interventions: Drug: Sertraline; Drug: Brexpiprazole Matching Placebo; Drug: Sertraline Matching Placebo
- Placebo (Placebo Comparator): Participants received oral brexpiprazole matching placebo tablet and oral sertraline matching placebo capsules up to Week 12.
  Interventions: Drug: Brexpiprazole Matching Placebo; Drug: Sertraline Matching Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole oral tablets.
  Other Names: OPC-34712; OPC-331
  Arms: Brexpiprazole; Brexpiprazole + Sertraline
Drug: Sertraline — Sertraline oral capsules.
  Other Names: Zoloft
  Arms: Brexpiprazole + Sertraline; Sertraline
Drug: Brexpiprazole Matching Placebo — Brexpiprazole matching placebo oral tablets.
  Arms: Placebo; Sertraline
Drug: Sertraline Matching Placebo — Sertraline matching placebo oral capsules.

SUMMARY:
To evaluate the safety, efficacy and tolerability of brexpiprazole (with placebo) as monotherapy or combination therapy with Zoloft (sertraline) in adults with PTSD.

DETAILED DESCRIPTION:
This trial is designed to assess the efficacy, safety and tolerability of flexible dose brexpiprazole as monotherapy or as combination therapy with Zoloft (Sertraline) in adult participants with PTSD.

This study will consist of a continuous 12-week, double-blind treatment period with a 14-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the years of 18-65 with a diagnosis of PTSD (diagnosis can be made at screening)

Exclusion Criteria:

* Index trauma event >15 years before screening
* Index trauma event at age <16
* Any traumatic event within 3 months of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - Investigational Site, Tuscaloosa, Alabama
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Rogers, Arkansas
  - Investigational Site, Bellflower, California
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Glendale, California
  - Investigational Site, National City, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Orange, California
  - Investigational Site, Redlands, California
  - Investigational Site, Riverside, California
  - Investigational Site, San Diego, California
  - Investigational Site, San Marcos, California
  - Investigational Site, Torrance, California
  - Investigational Site, Colorado Springs, Colorado
  - Investigational Site, Bradenton, Florida
  - Investigational Site, Fort Lauderdale, Florida
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Gainesville, Florida
  - Investigational Site, Jacksonville, Florida
  - Investigational Site, North Miami, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Decatur, Georgia
  - Investigational Site, Roswell, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Berlin, New Jersey
  - Investigational Site, Princeton, New Jersey
  - Investigational Site, Brooklyn, New York
  - Investigational Site, Cedarhurst, New York
  - Investigational Site, New York, New York
  - Investigational Site, Rochester, New York
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Raleigh, North Carolina
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Portland, Oregon
  - Investigational Site, Salem, Oregon
  - Investigational Site, Media, Pennsylvania
  - Investigational Site, Norristown, Pennsylvania
  - Investigational Site, Lincoln, Rhode Island
  - Investigational Site, Charleston, South Carolina
  - Investigational Site, Memphis, Tennessee
  - Investigational Site, Bellaire, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Wichita Falls, Texas
  - Investigational Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Hobart M, Chang D, Hefting N, Davis LL. Brexpiprazole in Combination With Sertraline and as Monotherapy in Posttraumatic Stress Disorder: A Full-Factorial Randomized Clinical Trial. J Clin Psychiatry. 2025 Feb 19;86(1):24m15577. doi: 10.4088/JCP.24m15577. PMID 40009045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 48 investigative sites in the United States from 26 January 2017 to 12 November 2018.
Pre-assignment Details: Of the 336 participants enrolled in the study, 321 participants diagnosed with post-traumatic stress disorder (PTSD) were randomized in 1:1:1:1 ratio to receive brexpiprazole monotherapy, brexpiprazole plus sertraline combination therapy, sertraline monotherapy or placebo up to Week 12.
Period: Overall Study
Arm/Group | Brexpiprazole + Sertraline | Brexpiprazole | Sertraline | Placebo
Started | 82 | 75 | 81 | 83
Safety Sample (Safety Sample included all participants who were randomized into this trial and were administered at least one dose of double-blind investigational medicinal product (IMP).) | 80 | 75 | 79 | 82
Intent to Treat (ITT) Sample (ITT Sample included all participants who were randomized in the trial and took at least one dose of double-blind IMP and have a Baseline and at least one post Baseline evaluation for the clinician-administered PTSD scale for diagnostic and statistical manual of mental disorders, 5th edition (DSM-5) CAPS-5 total score.) | 79 | 72 | 77 | 80
Completed | 58 | 50 | 59 | 64
Not Completed | 24 | 25 | 22 | 19
Not completed — Adverse Event | 6 | 7 | 4 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 6 | 5 | 5 | 6
Not completed — Non-Compliance With Study Drug | 1 | 1 | 1 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 10 | 11 | 6
Not completed — Withdrawal By Caregiver | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Sample included all participants randomized into this trial.
Groups:
- Brexpiprazole + Sertraline: Participants were administered oral brexpiprazole initial dose of 0.5 mg/day plus sertraline initial dose of 50 mg/day. The dose was up titrated to brexpiprazole maximum dose of 3 mg/day and sertraline maximum dose of 200 mg/day and continued thereafter up to Week 12 based on efficacy and tolerability. No dose reductions were allowed after Week 6 and no dose increments were allowed after Week 4. Participants also received sertraline matching placebo based on dose titration/adjustment up to Week 12.
- Placebo: Participants received oral brexpiprazole matching placebo tablet and oral sertraline matching placebo capsules up to Week12.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole + Sertraline | Brexpiprazole | Sertraline | Placebo | Total
Number analyzed (Participants) | 82 | 75 | 81 | 83 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.9) | 39.3 (10.6) | 38.6 (10.9) | 40.3 (11.0) | 39.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 51 | 48 | 199
  Male | 31 | 26 | 30 | 35 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 1 | 0 | 2 | 4
  Race: Asian | 1 | 2 | 0 | 1 | 4
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Race: Black or African American | 21 | 23 | 22 | 26 | 92
  Race: White | 55 | 43 | 53 | 46 | 197
  Race: Other | 3 | 5 | 6 | 8 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 13 | 11 | 11 | 14 | 49
  Ethnicity: Not Hispanic or Latino | 68 | 64 | 70 | 69 | 271
  Ethnicity: Other | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 75 | 81 | 83 | 321

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered Post-traumatic Stress Disorder (PTSD) Scale for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (CAPS-5) Total Score
Description: CAPS-5:clinician-rated, structured interview to assess PTSD diagnostic status, symptoms severity as defined by DSM-5. CAPS-5 Past Week version of scale was completed at Baseline and at all visits after Baseline. CAPS-5 was calculated by summing severity scores for 20 DSM-5 PTSD symptoms (items 1-20) from categories: Category B:Intrusion symptoms (5 items); Category C:Avoidance symptoms (2 items); Category D:Cognition and mood symptoms (7 items); Category E:Arousal and reactivity symptoms (6 items). CAPS-5 total score was imputed by adding all subscores from categories B,C,D,E. Each symptom was scored 0 (Absent) to 4 (Extreme/incapacitating), to yield a score with range 0-80. Higher scores=worse outcome. Mixed model repeated measure (MMRM) was used for analysis.
Time Frame: Baseline, Week 12
Population: ITT Sample included all participants who were randomized in the trial and took at least one dose of double-blind investigational medicinal product (IMP) and have a Baseline and at least one post Baseline evaluation for the CAPS-5 total score. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole + Sertraline | Brexpiprazole | Sertraline | Placebo
Number analyzed (Participants) | 59 | 48 | 58 | 62
score on a scale | -16.4 (1.43) | -12.2 (1.57) | -11.4 (1.46) | -10.5 (1.40)
Statistical Analysis 1: Comparison: Brexpiprazole + Sertraline vs Placebo; MMRM analysis with an unstructured (UN) variance covariance structure was performed. The model included fixed class-effect terms for treatment, trial site, type of trauma (combat related Yes/No), visit week, and an interaction term of treatment by visit week and included the interaction term of baseline values of CAPS-5 total score by visit week as a covariate; Test type: Superiority; p = 0.0021, Mixed Model Repeated Measures (MMRM); Least Squares (LS ) Mean Difference = -5.99, 95% CI 2-sided [-9.79 to -2.19]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; MMRM analysis with an UN variance covariance structure was performed. The model included fixed class-effect terms for treatment, trial site, type of trauma (combat related Yes/No), visit week, and an interaction term of treatment by visit week and included the interaction term of baseline values of CAPS-5 total score by visit week as a covariate; Test type: Superiority; p = 0.3868, MMRM; LS Mean Difference = -1.74, 95% CI 2-sided [-5.70 to 2.22]
Statistical Analysis 3: Comparison: Sertraline vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.6399, MMRM; LS Mean Difference = -0.91, 95% CI 2-sided [-4.74 to 2.92]
Statistical Analysis 4: Comparison: Brexpiprazole + Sertraline vs Sertraline; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0106, MMRM; LS Mean Difference = -5.08, 95% CI 2-sided [-8.96 to -1.20]
Statistical Analysis 5: Comparison: Brexpiprazole + Sertraline vs Brexpiprazole; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0384, MMRM; LS Mean Difference = -4.24, 95% CI 2-sided [-8.26 to -0.23]

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to 14 days after the last dose (Up to Week 14)
Description: Safety Sample included all participants who were randomized into this trial and were administered at least one dose of double-blind IMP.
Arm/Group | Brexpiprazole + Sertraline | Brexpiprazole | Sertraline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/75 | 0/79 | 1/82
Serious Adverse Events (participants affected / at risk) | 2/80 | 1/75 | 0/79 | 4/82
Other Adverse Events (participants affected / at risk) | 47/80 | 42/75 | 46/79 | 43/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + Sertraline (N=80) | Brexpiprazole (N=75) | Sertraline (N=79) | Placebo (N=82)
Chest pain (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + Sertraline (N=80) | Brexpiprazole (N=75) | Sertraline (N=79) | Placebo (N=82)
Constipation (Gastrointestinal disorders) | 4 | 2 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 7 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 6 | 10 | 7
Nausea (Gastrointestinal disorders) | 4 | 1 | 16 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Fatigue (General disorders) | 2 | 6 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 7 | 7
Weight increase (Investigations) | 10 | 6 | 1 | 7
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5 | 1 | 1
Akathisia (Nervous system disorders) | 5 | 10 | 3 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 5 | 5
Headache (Nervous system disorders) | 6 | 4 | 7 | 7
Sedation (Nervous system disorders) | 3 | 5 | 0 | 0
Somnolence (Nervous system disorders) | 8 | 5 | 3 | 7
Anorgasmia (Psychiatric disorders) | 4 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 4 | 0 | 4
Insomnia (Psychiatric disorders) | 2 | 5 | 4 | 3
Irritability (Psychiatric disorders) | 3 | 1 | 4 | 3
Delayed ejaculation (Reproductive system and breast disorders) | 4 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03033069/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT03033069/SAP_001.pdf